CLINICAL TRIAL: NCT03418324
Title: A Phase 2 Study of TRC105 (Anti-endoglin Antibody) With Abiraterone and With Enzalutamide in Metastatic, Castration Resistant Prostate Cancer Patients Progressing on Therapy
Brief Title: Study of TRC105 With Abiraterone and With Enzalutamide in Prostate Cancer Patients Progressing on Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Edwin Posadas, MD, Medical Director, Urologic Oncology Program, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2016-16-POSADAS-TRC105
Record Dates: First submitted 2018-01-23; First posted 2018-02-01 (Actual); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Metastatic Prostate Cancer; Castration Resistant Prostate Cancer; Metastatic Castration Resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carotuximab; abiraterone; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Intervention Model Description: Bayesian design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: TRC105 + Abiraterone (Experimental): Patients progressing on Abiraterone will undergo a washout period and then continue treatment with TRC105 + Abiraterone
  Interventions: Drug: TRC105; Drug: Abiraterone
- Arm E: TRC105 + Enzalutamide (Experimental): Patients progressing on Enzalutamide will undergo a washout period and then continue treatment with TRC105 + Enzalutamide
  Interventions: Drug: TRC105; Drug: Enzalutamide

INTERVENTIONS:
Drug: TRC105 — Patients will receive TRC105 10mg weekly x 4, and then 15 mg/kg every 2 weeks
  Other Names: Carotuximab
Drug: Abiraterone — Patients who are progressing on Abiraterone will undergo a washout period and then continue treatment with standard dosing of Abiraterone plus TRC105.
  Other Names: Zytiga
  Arms: Arm A: TRC105 + Abiraterone
Drug: Enzalutamide — Patients who are progressing on Enzalutamide will undergo a washout period and then continue standard treatment with Enzalutamide plus TRC105.
  Other Names: Xtandi
  Arms: Arm E: TRC105 + Enzalutamide

SUMMARY:
This research study is being done to measure the clinical benefit of TRC105 in combination with abiraterone or enzalutamide in metastatic, castration-resistant prostate cancer patients who are taking either abiraterone or enzalutamide and showing signs of biochemical progression without radiographic progression. A patient who is progressing on AR-therapy will continue the same AR-therapy on study with the addition of TRC105. The two arms will accrue in parallel and independently.

DETAILED DESCRIPTION:
This is a Phase II, open-label study of TRC105 (anti-endoglin antibody) in combination with abiraterone or enzalutamide in metastatic, castration-resistant prostate cancer patients who are taking either abiraterone or enzalutamide and showing signs of biochemical progression without radiographic progression. A patient who is progressing on AR-therapy will continue the same AR-therapy on study with the addition of TRC105. The two arms will accrue in parallel and independently.

There will be a 2-week washout of the active AR-targeted therapy prior to initiation of combination therapy. Tumor response should be assessed at a frequency of 8 weeks by CT/MRI chest, abdomen and pelvis as well as bone scan. Patients may continue on therapy until radiographic progression by RECIST 1.1 or PCWG3 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. History of metastatic, castration-resistant prostate cancer with rising PSA on either abiraterone or enzalutamide

   * PSA rise will be defined as an increase in PSA of 0.2 ng/mL or higher on at least 2 separate occasions greater than 1 week apart while on either abiraterone or enzalutamide
   * If there is a drop in serum PSA after the first rise, and the patient has another PSA rise which is greater than the first, the patient will still be considered eligible.
2. ECOG 0-2
3. Resolution of adverse events results as described below.

   * Laboratory abnormalities must meet values specified below in criteria #4
   * If the patient's most recent line of therapy is treatment with abiraterone or enzalutamide, then all adverse events must be resolved to Grade 2 or better
   * If the most recent line of therapy is any other treatment for mCRPC then all Adverse events must be resolved to grade 1 or better, with the exception of fatigue, alopecia and neuropathy (which must resolve to CTCAE grade 2)
4. Adequate organ function defined by:

   * AST and ALT < 2.5 x ULN
   * Total serum bilirubin < 1.5 x ULN
   * Platelets > 60,000
   * Hgb > 8.5 g/dL
   * Serum Cr <1.5 x ULN or a creatinine clearance > 30.
   * INR ≤ 1.2 unless the patient is receiving a direct Factor Xa inhibitor or a direct thrombin inhibitor
5. Patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate. Abstinence from intercourse is an acceptable form of contraception.

Exclusion Criteria:

1. Non-PSA producing prostate cancers- such as small cell prostate cancers or those prostate cancers which exhibit radiographic progression without PSA rise
2. Inability to tolerate standard doses of abiraterone (1000 mg daily) or enzalutamide (160 mg daily).
3. Other prior malignancy requiring active anticancer therapy
4. Prior exposure to TRC105 or any CD105 targeted antibody
5. Any major surgical procedure within 2 weeks of starting therapy
6. Uncontrolled chronic hypertension defined as sustained by systolic pressure (SBP) >150 mmHg or diastolic pressure (DBP) >90 despite optimal therapy.
7. Active bleeding or pathologic conditions that carries a high bleeding risk
8. Use of thrombolytics within 10 days prior to the first day of TRC105
9. Known hypersensitivity to Chinese hamster ovary products or other recombinant human, chimeric, or humanized antibodies
10. A known diagnosis of Osler-Weber-Rendu syndrome
11. Ascites or pericardial or pleural effusion requiring external drainage procedures
12. History of untreated brain involvement with cancer, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been administered for at least 28 days. Imaging for CNS disease will not be required for screening unless there is a history of a neurological finding such as new onset weakness or numbness that cannot be explained by other medical history.
13. Acute cardiovascular event within the past 6 months. An acute cardiovascular event will be defined as a myocardial infraction, NYHA Class II or worse congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), or CABG. Deep venous thrombosis within 6 months, unless the patient is anti-coagulated without the use of warfarin for at least 2 weeks. In this situation, low molecular weight heparin is preferred.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD FACP, Principal Investigator — Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to accrual February 5, 2018 and the first patient on study March 5, 2018. As of November 6, 2019, 12 patients have been consented, 11 were enrolled, and 11 were off-treatment and off-study. Study closed to accrual on May 1, 2019, as drug manufacturer has limited drug supply without plans to increase production.
Pre-assignment Details: Early accrual closure due to manufacturer's limited drug supply.
Period: Overall Study
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Started | 3 | 8
Completed | 2 | 6
Not Completed | 1 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide | Total
Number analyzed (Participants) | 2 | 6 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 2 | 4 | 6
Age, Continuous [Median (Full Range); unit: years] | 76.5 [74 to 79] | 72 [57 to 73] | 72 [57 to 79]
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (3.53) | 67.83 (6.97) | 70 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 6 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Benefit
Description: Number of participants with stabilization of disease for at least 2 months or disease improvement at any time from start of combination therapy by radiographic and/or biochemical criteria through treatment completion up to an estimated period of 24 months
  * radiographic improvement defined as a PR (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum. There can be no appearance of new lesions) or CR (Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions) by RECIST 1.1 or improvement by PCWG3 criteria
  * Biochemical response will be defined by PCWG3 criteria
  * Stabilization will be defined as the absence of progression by BOTH radiographic and biochemical criteria
Time Frame: Through study completion, average 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants
  Overall Clinical Benefit | 1 | 4
  Radiographic Improvement | 1 | 2
  Biochemical Response | 1 | 1
  Stabilization | 1 | 3
Statistical Analysis 1: Comparison: Arm A: TRC105 + Abiraterone; For this study, we are not comparing outcome measures between the two arms; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 50, 95% CI 2-sided [1.3 to 98.7] — Estimated values reflects the percentage of participants with overall clinical benefit
Statistical Analysis 2: Comparison: Arm E: TRC105 + Enzalutamide; For this study, we are not comparing outcome measures between the two groups; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 66.7, 95% CI 2-sided [22.3 to 95.7] — Estimated values reflects the percentage of participants with overall clinical benefit

2. Secondary Outcome: Adverse Events From TRC105 and Abiraterone or Enzalutamide
Description: Number of participants with grade 3/4 Adverse Events Related to investigational therapy as assessed Using CTCAE (v.4) up to 4 months from treatment initiation.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants
  Grade 3 | 1 | 1
  Grade 4 | 0 | 0

3. Secondary Outcome: Progression Free Survival
Description: Time (in Months) from treatment initiation to radiographic and clinical progression over study duration (estimated 24 months)
  - radiographic criteria measured by RECIST 1.1 [Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions plus an absolute increase of at least 5 mm, taking as reference the smallest sum recorded since the start of study]
Time Frame: 24 months
Population: Median progression free survival (months) (95% confidence interval). Not enough data (insufficient number of participants with events) to establish upper limit.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
months | 1.64 [1.64 to NA] — Not enough data (insufficient number of participants with events) to establish upper limit. | 4.46 [1.71 to NA] — Not enough data (insufficient number of participants with events) to establish upper limit.

4. Secondary Outcome: Clinical Benefit at Two Months
Description: Proportion of participants with stabilization of disease for two months or disease improvement at anytime from start of combination therapy to two months by radiographic and/or biochemical criteria
  * radiographic improvement defined as a PR (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum. There can be no appearance of new lesions) or CR (Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions) by RECIST 1.1 or improvement by PCWG3 criteria
  * Biochemical response will be defined by PCWG3 criteria
  * Stabilization will be defined as the absence of progression by BOTH radiographic and biochemical criteria
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants
  Clinical Benefit | 1 | 4
  Radiographic Improvement | 1 | 1
  Biochemical Response | 1 | 1
  Stabilization | 1 | 3
Statistical Analysis 1: Comparison: Arm A: TRC105 + Abiraterone; For this study, we are not comparing outcome measures between the two arms; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 50, 95% CI 2-sided [1.3 to 98.7]
Statistical Analysis 2: Comparison: Arm E: TRC105 + Enzalutamide; For this study, we are not comparing outcome measures between the two arms; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 66.7, 95% CI 2-sided [22.3 to 95.7]

5. Secondary Outcome: Clinical Benefit at Four Months
Description: Proportion of participants with stabilization of disease for at least 4 months or disease improvement at anytime from start of combination therapy to four months by radiographic and/or biochemical criteria
  * radiographic improvement defined as a PR (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum. There can be no appearance of new lesions) or CR (Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions) by RECIST 1.1 or improvement by PCWG3 criteria
  * Biochemical response will be defined by PCWG3 criteria
  * Stabilization will be defined as the absence of progression by BOTH radiographic and biochemical criteria
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants
  Clinical Benefit | 1 | 3
  Radiographic Improvement | 1 | 2
  Biochemical Response | 1 | 1
  Stabilization | 1 | 2
Statistical Analysis 1: Comparison: Arm A: TRC105 + Abiraterone; For this study, we are not comparing outcome measures between the two arms; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 50, 95% CI 2-sided [1.3 to 98.7]
Statistical Analysis 2: Comparison: Arm E: TRC105 + Enzalutamide; For this study, we are not comparing outcome measures between the two arms; Test type: Other — Binomial proportion (Clopper-Pearson exact confidence interval) for each arm; Binomial proportion = 50, 95% CI 2-sided [11.8 to 88.2]

6. Secondary Outcome: Clinical Benefit From PSA Serum Concentration (2 Months)
Description: Proportion of participants with stabilization of disease based on PSA serum concentration levels. Stabilization of disease refers to PSA values that do not meet criteria for progression where progression will be defined as a rise in serum PSA that is ≥ 25% and 2 ng/mL above nadir which is confirmed by a second value ≥ 3 weeks later.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants | 1 | 4

7. Secondary Outcome: Clinical Benefit From PSA Serum Concentration (4 Months)
Description: as for outcome 6
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
Number analyzed (Participants) | 2 | 6
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: 2 years
Description: 3 patients consented to Arm A, but only 2 were considered evaluable (1 patient considered unevaluable per physician decision prior to treatment start). 8 patients consented to Arm E, but 6 were considered evaluable. Of the 2 patients not included in Arm E, 1 patient was deemed unevaluable by physician decision prior to starting study treatment, and the other died prior to starting study treatment. Therefore, this number is reflected in All-Cause Mortality, and differs from SAEs and Other.
Arm/Group | Arm A: TRC105 + Abiraterone | Arm E: TRC105 + Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/8
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/6
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: TRC105 + Abiraterone (N=2) | Arm E: TRC105 + Enzalutamide (N=6)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cellulitis (peri-mandibular) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: TRC105 + Abiraterone (N=2) | Arm E: TRC105 + Enzalutamide (N=6)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Anemia Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2 (7) | 2 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 6 (10)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 1 (2) | 2 (2)
Generalized weakness (General disorders) | 1 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 2 (3) | 5 (6)
Guaiac + Stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Petechiae (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (3)
Cauda equina (Nervous system disorders) | 1 (1) | 0 (0)
Cellulitis (peri-mandibular) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Right leg sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Geographic Tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 2 (2)
MRSA (Infections and infestations) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Redness sclera left eye (Eye disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Vision decrease (binocular) (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early accrual closure due to manufacturer's limited drug supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03418324/Prot_SAP_000.pdf